CLINICAL TRIAL: NCT06865417
Title: A Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Filgotinib, With Single Arm Induction and Maintenance, in Pediatric Subjects (8 to <18 Years of Age) With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study Evaluating the Effects of Filgotinib in Children and Teenagers With Ulcerative Colitis
Acronym: Galapeduca
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-331
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Filgotinib (Experimental): Filgotinib
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — IP will be provided as commercially developed film-coated tablets (100 and 200 mg strength) or reduced-strength (65 mg) age-appropriate film-coated tablets for use in pediatric subjects aged at least 8 years and needs to be taken orally q.d. at approximately the same time every morning (with or without food).

SUMMARY:
The aim of this study is to evaluate the efficacy, safety, tolerability, and pharmacokinetics (PK) of filgotinib as a treatment for UC in children and adolescents aged from 8 to less than 18 years.

Approximately 80 subjects from 8 to <18 years of age with moderately to severely active UC, including a minimum of 8 subjects from 8 to <12 years of age, will be enrolled in this study.

During the study, eligible subjects will take the investigational product (IP) on-site at Week 4, Week 10, and Week 22 (in the morning; with or without food). On all other days, subjects will take IP at home (in the morning; with or without food).

Subjects who do not achieve mMCS remission and/or MCS response at Week 10 will continue with induction treatment until Week 22. Subjects who do not achieve PUCAI remission at Week 22 will be permanently discontinued from the study.

Subjects will all receive a filgotinib dose targeting the same systemic exposure as that observed in adults with UC treated with 200 mg q.d.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a minimum body weight (BW) of 15 kg.
* Subject:

  * has documented diagnosis of UC with a minimum duration of 3 months,
  * has mMCS of 5 to 9, and an MCS endoscopic score >=2, rectal bleeding >=1, and stool frequency >=1,
  * has had an inadequate response, loss of response, intolerance, or has medical contraindications to corticosteroids, immunosuppressants, and/or biologic therapy. This includes subjects who depend on corticosteroids to control their symptoms and who experience worsening of their disease when attempting to wean off corticosteroids.

Exclusion Criteria:

* Subject has a diagnosis of inflammatory bowel disease -unclassified or indeterminate colitis, isolated proctitis, or toxic megacolon.
* Subject has an active infection.
* Subject with a history of complicated herpes zoster infection (with multi-dermatomal, disseminated, ophthalmic, or central nervous system involvement).
* Currently on any therapy for chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex, herpes zoster, or atypical mycobacteria).
* Subject has a history of colectomy or extensive small bowel resection.
* Subject with psychological or cognitive difficulties that might interfere with study participation.
* Subject has any previous exposure to a Janus kinase inhibitor or medication with a similar mode of action (e.g. tofacitinib, baricitinib, upadacitinib).
* Female subject is pregnant or breast feeding or intending to become pregnant or breastfeed during the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of filgotinib in induction of remission and maintenance of effect in pediatric subjects with ulcerative colitis (UC) | Week 10
  Proportion of subjects achieving clinical remission based on modified Mayo Clinical Score (mMCS)
subjects with ulcerative colitis (UC) | Week 58
  Proportion of subjects achieving clinical remission based on mMCS

SECONDARY OUTCOMES:
Safety and tolerability of filgotinib in pediatric subjects with UC | Week 62
  Incidence of treatment-emergent adverse events (TEAEs), adverse events of interest, and laboratory abnormalities through follow-up
Safety and tolerability of filgotinib in pediatric subjects with UC | Week 58
  Change from baseline in body mass index (BMI)
Safety and tolerability of filgotinib in pediatric subjects with U | Week 58
  Change from baseline in height velocity

CONTACTS AND LOCATIONS:
Locations (51):
- Belgium (3):
  - Association Hospitaliere De Bruxelles Hopital Universitaire Des Enfants Reine Fabiola, Brussels, Brussels Capital
  - Centre Hospitalier Regional De La Citadelle, Liège, Liege
  - Centre Hospitalier Universitaire Dinant Godinne Sainte-Elisabeth-UCL-Namur, Namur, Namur
- Croatia (3):
  - Klinicki Bolnicki Centar Osijek, Osijek, Croatia
  - Children's Hospital Zagreb, Zagreb, Croatia
  - University Hospital Centre Zagreb, Zagreb, Croatia
- France (6):
  - Hospital Femme Mere Enfant, Bron, France
  - Centre Hospitalier Universitaire De Dijon, Dijon, France
  - Hopital Saint Vincent de Paul - GHICL Lille, Lille, France
  - CHU de Montpellier, Montpellier, France
  - Centre Hospitalier Universitaire De Rennes, Rennes, France
  - Centre Hospitalier Regional Universitaire De Tours, Tours, France
- Germany (4):
  - Universitaetsklinikum Aachen AöR, Aachen, Germany
  - Universitaetsklinikum Leipzig AöR, Leipzig, Germany
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Mainz, Germany
  - Universitaetsklinikum Tuebingen AöR, Tübingen, Germany
- Greece (4):
  - Athens General Children's Hospital Panagioti And Aglaia Kyriakou, Athens, Greece
  - University General Hospital Attikon, Athens, Greece
  - General Hospital Of Thessaloniki Papageorgiou, Efkarpia, Greece
  - Hippokration Hospital, Thessaloniki, Greece
- Children's Health Ireland, Dublin, Ireland, Ireland
- Italy (7):
  - Azienda Ospedaliero-Universitaria Ss Antonio E Biagio E Cesare Arrigo, Alessandria, Italy
  - Azienda Ospedaliero Universitaria dell Marche I G M Lancisi G Salesi, Ancona, Italy
  - ASST Fatebenefratelli Sacco, Milan, Italy
  - Azienda Ospedaliera Universitaria Federico II Di Napoli, Naples, Italy
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Rome, Italy
  - Ospedale Pediatrico Bambino Gesu, Rome, Italy
  - IRCCS Materno Infantile Burlo Garofolo, Trieste, Italy
- Norway (2):
  - Oslo University Hospital HF, Oslo, Norway
  - Sykehuset I Vestfold HF, Tønsberg, Norway
- Poland (6):
  - In Vivo Sp. z o.o., Bydgoszcz, Poland
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk, Poland
  - Uniwersytecki Szpital Dzieciecy W Krakowie, Krakow, Poland
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Poland
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów, Poland
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Poland
- Portugal (3):
  - CCAB Centro Clinico Academico Braga Associacao, Braga, Portugal
  - Hospital Pediátrico de Coimbra, Coimbra, Portugal
  - Unidade Local De Saude Do Alto Minho E.P.E., Viana do Castelo, Portugal
- Romania (2):
  - Dr. Victor Gomoiu Clinical Children Hospital, Bucharest, Romania
  - Spitalul Clinic De Urgenta Pentru Copii Louis Turcanu Timisoara, Timișoara, Romania
- Spain (2):
  - Hospital Germans Trias I Pujol, Badalona, Spain
  - Hospital Universitario Reina Sofia, Córdoba, Spain
- United Kingdom (8):
  - Bristol Royal Infirmary, Bristol
  - Noah's Ark Children's Hospital, Cardiff
  - Ninewells Hospital, Glasgow
  - Alder Hey Children's Hospital, Liverpool
  - Chelsea and Westminster Hospital, London
  - The Newcastle upon Tyne Hospital FT, Newcastle
  - John Radcliffe Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield